CLINICAL TRIAL: NCT02851732
Title: A Cluster Randomized Trial Evaluating the Effect of a Multifaceted Intervention to Increase Evidence Based Strategies Usage for Cardiovascular Prevention.
Brief Title: Brazilian inteRvention to Increase eviDence usaGe in practicE - Cardiovascular Prevention
Acronym: BRIDGE-CV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Instituto de Pesquisa, Otavio Berwanger, Hospital do Coracao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BRIDGE0003
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases
Keywords: Quality Improvement; Cluster Analysis
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Clusters randomized to the control group will keep their usual practice standards. Patient screening will be performed at the outpatient clinics and primary care centers. Both groups must complete the following forms: "Admission", "06 months", and "12 months". Data collection will be performed from medical records by an independent professional not involved in patient care. Furthermore, study coordinator and data collectors from the sites, when asked, must provide appropriate documents for adjudication purposes.
- Intervention (Experimental): Educational multifaceted intervention can increase the evidence based prescriptions. If this is the case, this tool package may be offered as a quality improvement intervention for all hospitals. Health care professionals from each institution one being a physician (acting as a local leader) and the other being a research nurse (acting as a case manager) must attend the training course for high cardiovascular risk patients that will take place at HCor.
  Interventions: Behavioral: Quality Improvement Intervention

INTERVENTIONS:
Behavioral: Quality Improvement Intervention — The quality improvement intervention includes case management, reminders, check lists, educational materials, and audit and feedback reports
  Arms: Intervention

SUMMARY:
The purpose of the study is assess the impact of a multifaceted quality improvement intervention in adherence to evidence based therapies prescription (according to local guidelines) for cardiovascular prevention in high risk patients in 12 months.

DETAILED DESCRIPTION:
The quality improvement strategy being assessed in this study will be applied to the healthcare team, thus any intervention that is not well established in the literature will not be prescribed to the patients. Thus, this trial does not imply any additional risk for patients.

Furthermore, if this strategy is proved to be effective, it may be offered as a new clinical practice that might benefit brazilian patients.

BRIDGE-CV consists of a quality improvement project by the incorporation of evidence based interventions in public and private hospitals in Brazil. The chosen setting is cardiovascular prevention in high risk patients since cardiovascular diseases represent the major cause of death in Brazil.

It will be developed a cluster randomized trial, where hospitals will be allocated to receive or not the multifaceted intervention.

The patients will be followed for 12 months in order to assess if the multifaceted intervention can increase the evidence based prescriptions. If this is the case, this tool package may be offered as a quality improvement intervention for all hospitals.

Sites will be selected through the HCor investigators network. Invited sites must complete a screening form in order to verify eligibility and feasibility of application of the BRIDGE CV tools.Clusters will be randomized and allocated 1:1 to the Multifaceted Intervention Group or to the Control Group. Once the hospital/center is allocated to one of the groups every patient at that institution must be assisted following the same procedures.

The randomization list will be created considering a random function with equal probability of being allocated to each of the groups. Each site will receive a code number and just this numbers will be used during randomization. This procedure will be performed by the HCor statistician ensuring allocation concealment. The study coordinator will inform the site what procedures must be taken, without revealing to the statistician which hospitals are allocated to the intervention group.

The sample will be stratified considering primary care centers and secondary/tertiary outpatients' clinics.

Considering the open nature of the study, treatment allocation will not be blinded to the investigators, health care providers and patients.

However, clinical outcomes will be assessed and validated by a blinded committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 40 years old, with manifested atherothrombotic diseases ( coronary artery disease, stroke or transient ischemic attack, or peripheral artery disease)

Exclusion Criteria:

* Patients from institutions that don't provide the Institutional Authorization Term, as well as patients that withdraw Inform Consent for Data Collection.
* Patients with a history of atrial fibrillation or that at the discretion of the physician needs anticoagulation, will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1623 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Adherence to evidence based therapies | 12 months
  Adherence to evidence based therapies ( aspirin/antiplatelets , lipid lowering agents(statins) and ACE inhibitors/ARB) in an "all or none" model for patients without contra indication in a period of 12 months.

SECONDARY OUTCOMES:
Adherence to evidence based therapies | six and twelve months
  Adherence to aspirin/antiplatelets, lipid lowering agents(statins) and ACE Inhibitors/ARB in patients without contra indications (All or None Model).
LDL < 100mg/dL in 12 months | 12 months
  Percentage of eligible patients with LDL < 100mg/dL
LDL < 70mg/dL in 12 months | 12 months
  Percentage of eligible patients with LDL < 70mg/dL
Adherence to Lipid Lowering Agents (Statins) | 12 months
  Adherence to Lipid Lowering Agents (Statins) in patients without contraindications
Adherence to Antiplatelets | 12 months
  Adherence to Antiplatelets in Patients without contra-indications
Adherence to ACE inhibitors or ARBs | 12 Months
  Adherence to ACE inhibitors or ARBs in patients without contra-indications
Composite Outcome of Major Cardiovascular Events | 12 months
  Composite Outcome (death, non fatal myocardial infarction and non fatal stroke)
Adherence to Beta Blockers | 12 months
  Adherence to Beta Blockers in patients with a history of myocardial infarction and without contra-indications
Smoke Cessation Education | 12 Months
  Smoke Cessation Education delivered to smokers
Blood Pressure < 140 x 90 mmHg | 12 months
  Percentage of patients with blood pressure < 140 x 90 mmHg
Blood Pressure < 120 mmHg | 12 months
  Percentage of patients with blood pressure < 140 x 90 mmHg

REFERENCES:
- [Derived] Machline-Carrion MJ, Soares RM, Damiani LP, Campos VB, Sampaio B, Fonseca FH, Izar MC, Amodeo C, Pontes-Neto OM, Santos JY, Gomes SPDC, Saraiva JFK, Ramacciotti E, Barros E Silva PGM, Lopes RD, Brandao da Silva N, Guimaraes HP, Piegas L, Stein AT, Berwanger O; BRIDGE Cardiovascular Prevention Investigators. Effect of a Multifaceted Quality Improvement Intervention on the Prescription of Evidence-Based Treatment in Patients at High Cardiovascular Risk in Brazil: The BRIDGE Cardiovascular Prevention Cluster Randomized Clinical Trial. JAMA Cardiol. 2019 May 1;4(5):408-417. doi: 10.1001/jamacardio.2019.0649. PMID 30942842